CLINICAL TRIAL: NCT00615654
Title: A Randomized Clinical Trial of Aquatic Physiotherapy Program on Functional Capacity in Patients With Fibromyalgia.
Brief Title: Aquatic Physical Therapy in Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sao Camilo University Center (Other)
Responsible Party: Physiotherapy Department, Clinical School São Camilo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01; 01
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-01

CONDITIONS: Fibromyalgia
Keywords: Hydrotherapy,; RCT,
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Other)
  Interventions: Other: aquatic physical therapy

INTERVENTIONS:
Other: aquatic physical therapy — The aquatic physiotherapy program for the SG was applied twice a week, in groups of six to seven people, with sessions lasting 40 minutes, over a 12-week period. The Control Group protocol included maintenance of the individuals' medication therapy and absence of any physical activity during the study period.

SUMMARY:
Objective: To investigate whether patients undergoing aquatic physiotherapy in groups improve their functional capacity, by means of the distance covered in the six-minute walk test (6WT), and to compare this with a control group. Methods: Forty women that had not been practicing regular physical activity for one year were randomly allocated either to the Study Group (SG) to undergo an aquatic physiotherapy program in groups applied twice a week, including aerobic exercises, muscle strengthening and relaxation for 12 weeks, or to the Control Group (CG), which did not do any physical activity. Both groups maintained their treatment with medications. All patients underwent two evaluations: one at the start and the other after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with a medical diagnosis of FS, without age restrictions and without impaired cognition, who had not been practicing regular physical activity for one year

Exclusion Criteria:

* Presence of other rheumatic diseases and cardiovascular problems
* Smoking
* Absence of medical permission for swimming pool activities
* Starting other therapies, or changes to and/or discontinuation of medical treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
functional capacity | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela O Gimenes, Ms, Principal Investigator — São Camilo University Center
Locations (1):
- São Camilo University Center, São Paulo, São Paulo, Brazil